CLINICAL TRIAL: NCT01837290
Title: The Effect of Dexmedetomine Premedication on the Bispectral Index Values Using Sedation With Propofol During Spinal Anesthesia on Geriatric Chronic Renal Failure Patients Undergoing Hip Fracture Surgery The Effect of Dexmedetomine Premedication on the Bispectral Index Values Using Sedation With Propofol During Spinal Anesthesia on Geriatric Chronic Renal Failure Patients Undergoing Hip Fracture Surgery
Brief Title: Effects of Dexmedetomidine Premedication on Geriatric Patients With Chronic Renal Failure Undergoing Hip Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Pinar Ergenoglu, Specialist Doctor, Anesthesiology and Reanimation Department, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KA12/166
Record Dates: First submitted 2013-04-17; First posted 2013-04-23 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Renal Failure; Hip Fracture
Keywords: Renal failure,; hip fracture,; spinal anesthesia,; dexmedetomidine; patient
MeSH Terms: conditions — Kidney Failure, Chronic; Hip Fractures; Renal Insufficiency | interventions — Premedication; Dexmedetomidine; Midazolam; Sodium Chloride; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Dexmedetomidine (Group D) (Active Comparator): Midazolam 0.02 mg/kg intravenously + 0.5 μg/kg/10 min dexmedetomidine infusion for premedication + Spinal block (Hyperbaric bupivacaine 0.5% 12.5 mg) (n=30)
  Interventions: Drug: dexmedetomidine infusion for premedication; Drug: Midazolam; Drug: Spinal block with hyperbaric bupivacaine 0.5% 12.5 mg
- Group Control (Group C) (Placebo Comparator): Midazolam 0.02 mg/kg + saline infusion for premedication; Spinal block (Hyperbaric bupivacaine 0.5% 12.5mg) (n=30)
  Interventions: Drug: Midazolam; Drug: saline infusion; Drug: Spinal block with hyperbaric bupivacaine 0.5% 12.5 mg

INTERVENTIONS:
Drug: dexmedetomidine infusion for premedication — Group Dexmedetomidine (Group D): Midazolam 0.02 mg/kg + 0.5 μg/kg/10 min dexmedetomidine infusion for premedication; Spinal block (Hyperbaric bupivacaine 0.5% 12.5 mg) (n=30)
  Other Names: Precedex 200mcg/2ml; 121/87; Hospira İnc., Rocky Mount, NC 27801 USA
  Arms: Group Dexmedetomidine (Group D)
Drug: Midazolam — intravenous Midazolam 0.02 mg/kg for premedication
  Other Names: Demizolam; Dem İlaç San. ve Tic AŞ.
Drug: saline infusion — Saline infusion to facilitate blinding
  Other Names: 0.9% sodium chloride solution
  Arms: Group Control (Group C)
Drug: Spinal block with hyperbaric bupivacaine 0.5% 12.5 mg — Hyperbaric bupivacaine injection for spinal block
  Other Names: Marcaine Spinal Heavy 0.5%; Astra Zeneca; 21.01.2000-194/86

SUMMARY:
Geriatric patients (age ≥ 65 years) undergo surgery for hip fractures that develops due to osteoporosis and falls. Dialysis-dependent chronic kidney disease is associated with an increased risk of cardiovascular comorbidity. Elective or urgent surgical operations may be required for geriatric patients with end stage renal disease. These patients have severe comorbidities, fluid, electrolyte disturbances and drug metabolism abnormalities during the perioperative period. For this reasons a careful anesthesia plan should be planned and performed. Spinal anesthesia can be used for hip fracture surgery at geriatric patients with chronic renal failure. Anterograde femoral intramedullary nailing can be performed in supine position with a fracture table. Intraoperative sedation might be necessary for patients under regional anesthesia on traction table. Dexmedetomidine is an alpha 2 receptor agonist that is being used as an agent for its sedative and adjuvant analgesic effects.

The aim of this study is to evaluate the effects of dexmedetomidine premedication on geriatric patients with end stage renal disease, who will be undergoing a surgical operation for hip fracture under spinal anesthesia with hyperbaric bupivacaine and BIS (Bispectral Index) guided sedation with intraoperative propofol infusion.

DETAILED DESCRIPTION:
Patients will be randomized into two separate groups.Group Dexmedetomidine (Group D): Midazolam 0.02 mg/kg + 0.5 μg/kg/10 min dexmedetomidine infusion for premedication; Spinal block (Hyperbaric bupivacaine 0.5% 12.5 mg) (n=30) Group Control (Group C): Midazolam 0.02 mg/kg + saline infusion for premedication; Spinal block (Hyperbaric bupivacaine 0.5% 12.5mg) (n=30)

In this randomized double-blinded study, drugs will be prepared by an anesthesia technician who is not part of the study. The patients will be monitored with a pulse-oxymeter, 5-channel ECG, noninvasive blood pressure and BIS at the preoperative preparation room. BIS monitoring electrodes will be placed on the forehead of the patient. Study drugs will be administered to the patient by another anesthesiologist who is also not taking part in the study at the preparation room preoperatively. Dexmedetomidine (0.5 μg/kg) in 20 ml saline will be administered in 10 minutes, with an infusion pump. An equivalent volume of saline solution will be given to the control group with same method. Baseline, 1., 3., 5., 10., minute BIS SpO2, systolic, diastolic and mean arteriel pressure values will be recorded. At this period 500 ml of 0.9% NaCl will be infused. The patient will then be transported to the operating room with the supervision of this anesthesiologist. The intraoperative and postoperative follow-up of the patients will be performed by another anesthesiologist who has been blinded to the study drugs as well as the group distribution. Routine anesthesia monitoring will be performed with pulse-oxymeter, 5-lead ECG, noninvasive blood pressure measurement, pulse oxymetry and BIS. Before induction of the spinal block basal systolic, diastolic and mean blood pressures, heart rate, peripheral oxygen saturation and BIS values will be recorded. Lumbar puncture will be performed in lateral decubitis position with a Quincke 27 gauge spinal needle at the L3-L4 interspaces using the midline approach. Patients will be promptly rotated supine position after block induction. Induction of the spinal block will be accepted as 0 for all intraoperative data recordings. Systolic, diastolic and mean blood pressures, heart rate, peripheral oxygen saturation and BIS values will be recorded at 1.,3. 5. minutes and every 5 minutes for the first hour and following that every 15 minutes during surgery.

Hypotension will be described as a drop off in systolic pressure by greater then 25% from the baseline or in case systolic blood pressure decreases below 90 mm Hg, 5 mg ephedrine will be administered intravenously and the rate of crystalloid infusion will be increased.

The sensorial block level and the motor block level will be tested with the pinprick test and Bromage scale (Bromage Scale; 0: No motor block: full flexion of knee and foot, 1: Inability to raise extended leg. Just able to move knee, 2: Inability to flex knee. Able to move foot only, 3: Inability to flex ankle joint. Unable to move foot or knee), respectively. Propofol infusion will be started in all patients at a dose of 50 mcg/kg/min after the level of block arises to T10 dermatome level. Target BIS values will be between 70 and 80. Infusion rate will be titrate to provide the targeted BIS levels.The time when BIS < 80 will be recorded. In case BIS<70, propofol infusion rate will be reduced. ''Observer's assessment of alertness/sedation (OAA/S)'' scale (OAAS score 5-awake and responds readily to name spoken in normal tone, OAAS score 4-lethargic responses to name in normal tone, OAAS score 3-responds only after name is called loudly and/or repeatedly, OAAS score 2-responds only after name called loudly and mild shaking, OAAS score 1-does not respond when name is called loudly and mild shaking or prodding, OAAS score 0-does not respond to noxious stimulation) will be used for evaluating the level of sedation, with a target of OAA/S ≤ 5. OAA/S scores will be registered at the same time points. Propofol infusion will be ended at the beginning of skin suturing, and BIS>90 time will be recorded.

Patients will be monitored at the postoperative care unit and all monitoring parameters (MAP, SAP, DAP, BIS, OASS) will be registered at every 5 minutes for one hour. Criteria for transferring the ward are BIS>90, OAA/S=5, Bromage=0-1 Duration of the surgery, the amount of bleeding, vasoactive drug need, the time necessary to reach the targeted level of sedation (BIS≤80), the amount of propofol infusion, propofol dose required for targeted BIS levels and the total propofol consumption recovery time (BIS>90) first analgesic requirement time (VAS: Visual Analogue Scale;0=no pain, 10=worst pain possible,VAS≥3) and the complications will be recorded. Side effects and possible complications during the intraoperative period and the postoperative follow-up include: hypotension (SBP<90 mmHg), bradycardia (CR < 60/min), hypoxia (SpO2≤ 94 %), nausea, vomiting, and respiratory depression will be recorded and the necessary medical interventions will be administered.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (above 65 years of age)
* end stage renal failure on dialysis treatment (Glomerular filtration rate <15, Stage 5)
* hip fracture

Exclusion Criteria:

* Patients with decompensated respiratory or heart failure,
* liver failure
* morbid obesity
* mental disorders
* cognitive disorders
* language problems
* patients with a contraindication for regional anesthesia (coagulopathy, history of anticoagulant use, spinal cord disease and patients who rejected spinal anesthesia)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Decrease at the propofol doses and postoperative early recovery | up to first 6 hours for postoperative pain management
  In addition patients will be followed postoperatively first 6 hours for postoperative pain management at the ward.

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof., MD, Study Director — Baskent University School of Medicine
Locations (3):
- Turkey (Türkiye) (3):
  - Baskent University School of Medicine Adana Research and Teaching Center, Adana
  - Baskent University School of Medicine Adana Teaching and Research Center, Adana
  - Baskent University School of Medicine Adana Teaching and Research Hospital, Adana

REFERENCES:
- [Background] Ozkan-Seyhan T, Sungur MO, Senturk E, Karadeniz M, Basel A, Senturk M, Akpir K. BIS guided sedation with propofol during spinal anaesthesia: influence of anaesthetic level on sedation requirement. Br J Anaesth. 2006 May;96(5):645-9. doi: 10.1093/bja/ael055. Epub 2006 Mar 10. PMID 16531442
- [Derived] Ergenoglu P, Akin S, Bali C, Eker HE, Yalcin Cok O, Aribogan A. Effect of low dose dexmedetomidine premedication on propofol consumption in geriatric end stage renal disease patients. Braz J Anesthesiol. 2015 Sep-Oct;65(5):326-32. doi: 10.1016/j.bjane.2014.11.002. Epub 2015 May 2. PMID 26323728